CLINICAL TRIAL: NCT02309398
Title: Improving Care for Cardiovascular Disease in China: A Collaborative Project of AHA and CSC (CCC Project) - Atrial Fibrillation
Brief Title: CCC Project - Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Collaborators: American Heart Association (Other); Chinese Society of Cardiology (Other)
Responsible Party: Principal Investigator, Dong ZHAO, Principal Investigator, Beijing Institute of Heart, Lung and Blood Vessel Diseases
Other Study IDs: CCC-AF-2014
Record Dates: First submitted 2014-11-30; First posted 2014-12-05 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to develop and implement quality improvement programs for the treatment of atrial fibrillation (AF) in China based on the successful experience of the AHA-Get with the Guidelines program. This program will use data collection, analysis, feedback, and process improvement to extend the use of evidence-based guidelines throughout the healthcare system and improve patient care of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with discharge diagnosis as atrial fibrillation in 150 tertiary and 100 secondary hospitals.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients of atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 67028 (Actual)
Dates: Start 2015-01; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
The overall composite of six performance measures for AF care | Duration of hospital stay, an expected average of 1 week
  Performance measures for AF care including:
  1. Proportion of patients received assessment of thromboembolic risk factors
  2. Proportion of patients discharged on warfarin or other anticoagulant drug
  3. Proportion of patients discharged on warfarin who have PT/INR follow-up planned prior to hospital discharge
  4. Proportion of patients with left ventricular systolic dysfunction prescribed an ACEI or ARB at hospital discharge
  5. Proportion of patients with left ventricular systolic dysfunction prescribed a beta blocker at hospital discharge
  6. Proportion of patients with either coronary artery disease, cerebrovascular accident/transient ischemic attack, peripheral vascular disease or diabetes who were prescribed a statin at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Dong Zhao, Ph. D, Principal Investigator — Beijing Institute of Heart, Lung and Blood Vessel Diseases
Locations (1):
- Beijing An Zhen Hospital, Beijing, China

REFERENCES:
- [Result] Hao Y, Liu J, Smith SC, Huo Y, Fonarow GC, Ge J, Liu J, Taubert KA, Morgan L, Guo Y, Zhou M, Zhao D, Ma C; CCC-AF Investigators. Rationale and design of the improving Care for Cardiovascular Disease in China (CCC) project: a national registry to improve management of atrial fibrillation. BMJ Open. 2018 Jul 5;8(7):e020968. doi: 10.1136/bmjopen-2017-020968. PMID 29980544
- [Derived] Han K, Li X, Fu B, Li M, Liu T, Peng Y, Liu J, Yang N, Hao Y, Jiang C, Tang R, Dong J, Zhao D, Long D, Ma C. Elevated Resting Heart Rate in Hospitalized Patients With Atrial Fibrillation Is Associated With Increased Cardiovascular Risk. Cardiovasc Ther. 2026 Jan 26;2026:2106637. doi: 10.1155/cdr/2106637. eCollection 2026. PMID 41608332
- [Derived] Tong XY, Lin J, Sun ZQ, He Q, Zhan Y, Jiang CX, Tang RB, Sang CH, Ning M, Jia CQ, Feng L, Wang W, Zhao X, Li CY, Li SN, Guo XY, Liu T, Li MM, Yang N, Hao YC, Liu J, Liu J, Xie J, Long DY, Dong JZ, Zhao D, Ma CS. Low-density lipoprotein cholesterol levels and in-hospital bleeding in patients with atrial fibrillation: findings from CCC-AF project. Front Cardiovasc Med. 2025 Jun 12;12:1574796. doi: 10.3389/fcvm.2025.1574796. eCollection 2025. PMID 40574812
- [Derived] Yang N, Sun Z, Liu J, Hao Y, Long D, Zhao D, Liu J; CCC-AF Investigators. Impact of insurance coverage for non-vitamin K antagonist oral anticoagulants on quality of care and care disparities in patients hospitalised with atrial fibrillation in tertiary hospitals in China: interrupted time series analysis. BMJ Open. 2025 Feb 22;15(2):e088539. doi: 10.1136/bmjopen-2024-088539. PMID 39986999
- [Derived] Xia Y, Jiang J, Fan F, Pan Y, Zhou J, Zhang Y, Li J, Liu J, Yang N, Hao Y, Zhao D, Liu J, Ma C, Huo Y; CCC-AF investigators. Prevalence, Characteristics, and Treatment Strategy of Different Types of Heart Failure in Patients With Nonvalvular Atrial Fibrillation. J Am Heart Assoc. 2024 Oct;13(19):e033941. doi: 10.1161/JAHA.123.033941. Epub 2024 Sep 30. PMID 39344652
- [Derived] Lin J, Long D, Jiang C, Sang C, Tang R, Li S, Wang W, Guo X, Ning M, Sun Z, Yang N, Hao Y, Liu J, Liu J, Du X, Morgan L, Fonarow GC, Smith SC Jr, Lip GYH, Zhao D, Dong J, Ma C; CCC-AF investigators. Oral anti-coagulants use in Chinese hospitalized patients with atrial fibrillation. Chin Med J (Engl). 2024 Jan 20;137(2):172-180. doi: 10.1097/CM9.0000000000002915. Epub 2023 Dec 22. PMID 38146256
- [Derived] He P, Pan Y, Jiang J, Fan F, Zhou J, Xia Y, Liu J, Yang N, Hao Y, Li J, Liu J, Zhao D, Huo Y; CCC-AF investigators. In-hospital therapies and determinants of treatment strategy selection in patients with atrial fibrillation and left ventricular systolic dysfunction in China: a retrospective study based on the Improving Care for Cardiovascular Disease in China-Atrial Fibrillation (CCC-AF) project, 2015-2019. BMJ Open. 2023 Jun 5;13(6):e070070. doi: 10.1136/bmjopen-2022-070070. PMID 37277219